CLINICAL TRIAL: NCT00528801
Title: Neuropsychological Dysfunction and Neuroimaging Abnormalities in Neurologically Intact Adults With Sickle Cell Disease
Brief Title: Examining Cognitive Function and Brain Abnormalities in Adults With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Elliott Vichinsky, Children's Hospital of Oakland and Research Institute
Other Study IDs: 480; U54HL070587 (NIH); U54HL070587-04 (NIH)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Hemoglobin SS; Hemoglobin SB0
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases (CLOSED): These are patients diagnosed with sickle cell disease (confirmed by hemoglobin electrophoresis).
  Interventions: Behavioral: NP Battery; Procedure: MRI
- Controls (CLOSED): These are persons that do not have sickle cell disease (confirmed by hemoglobin electrophoresis); matched to cases by age, gender, and education level
  Interventions: Behavioral: NP Battery; Procedure: MRI

INTERVENTIONS:
Behavioral: NP Battery — Neuropsych Battery with 7 different tests that evaluate the patients neurological functioning.
  Other Names: The Weschler Adult Intelligence Scale - Third Edition; The Woodcock Johnson Revised - Test of Achievement; The Delis-Kaplan Function System; The Wisconsin Card Sorting test; The Test of Everday Attention; The California Verbal Learning Test; The Weschler Memory Scales - Third Edition
Procedure: MRI — The MRI is a standard procedure involving 30 minutes under the machine in order to obtain various images of the patients brain.

SUMMARY:
Sickle cell disease (SCD), also known as sickle cell anemia, is an inherited blood disease that can cause intense pain episodes and may lead to organ failure. Preliminary studies have shown that adults with SCD may have brain abnormalities that contribute to problems with cognitive functioning, including attention and memory difficulties. This study will use brain magnetic resonance imaging (MRI) and neuropsychological testing to examine the differences in cognitive functioning in adults with SCD and adults without SCD.

212 subjects participated in this cross-sectional study consisting of screening questionnaires, a neuropsychological testing battery, and MRI testing. Enrollment into this study ended in May 2008.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder. Symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." In the past, SCD was considered a fatal disease, and many people with SCD died at a young age. Due to advances in medical care, people with SCD are now living longer lives; however, they often experience a deterioration in quality of life due to progressive organ failure. Past research has suggested that children with SCD commonly have frontal lobe dysfunction syndrome, which is a brain disorder that can affect cognitive functioning in areas such as attention, concentration, information processing, and decision making. Often times, however, neurocognitive and brain disorders are not diagnosed or treated in people with SCD. In preliminary brain imaging studies, at least half of adult participants with SCD had cognitive dysfunction that could be seen in images of the brain, while participants without SCD rarely had visible changes in the brain. Brain dysfunction may be one of the most important and least-studied problems affecting adults with SCD. The purpose of this study is to evaluate the extent of cognitive functioning problems in adults with SCD. The study will also determine if there is a connection between cognitive functioning problems and abnormalities seen on MRI brain images of adults with SCD.

This study is an observational case/control study that will enroll adults with SCD and a control group of healthy adults who do not have SCD. At a study visit on Day 1, participants will undergo blood collection and will complete psychosocial questionnaires. Female participants will provide a urine sample for pregnancy testing. Study researchers will conduct a medical record review, a physical exam, and a neurological exam. They will also interview participants to collect medical history information. On Day 2, participants will undergo either a brain MRI or neuropsychological testing; on Day 3, the other procedure will be completed. On Day 4, study researchers will explain the study procedure results to participants. Participants will be asked if they are willing to take part in a second phase of the study in the future. Enrollment into this study ended in May 2008.

A pilot interventional study follows this study, and is reported separately in ClinicalTrials.gov under NCT 00850018.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as cases into the study:

1. Adult between the ages of 21 and 55
2. African descent
3. Proficient/fluent in English
4. Hemoglobin electrophoresis confirming hemoglobin SS or SB0 (%A <= 15)
5. Hemoglobin <= 10 g/dL
6. Capable of giving informed consent for the protocol

Individuals who meet all of the following criteria are eligible for enrollment as community controls into the study:

1. Adult between the ages of 21 and 55
2. African descent
3. Proficient/fluent in English
4. Capable of giving informed consent for the protocol

Exclusion Criteria:

Individuals who meet any of the following criteria are disqualified from enrollment in the case group of the study:

1. Overt stroke
2. Previous evidence of an abnormal MRI or CT other than small peri-ventricular or watershed lesions
3. History of head injury that resulted in neurological symptoms or medical visit
4. Abnormal neurologic exam with focal findings
5. Mini-Mental Status Examination (MMSE) score of < 20
6. Profile of Mood States (POMS) score on the Depression-Dejection Subscale suggestive of a clinical depression (score > 40)
7. Alcohol consumption exceeding 14 drinks/week if female, 21 drinks/week if male
8. Drug abuse, defined as using non-prescribed medication
9. History of claustrophobia and/or presence of metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body
10. Pregnancy
11. Baseline blood pressure > 140/90 on two repeated measurements. A second measurement is needed only if the first is > 140/90
12. History of uncontrolled hypertension
13. Any chronic disorder that may result in neurocognitive or brain dysfunction that is not secondary to SCD including:

    1. Inflammatory arterial disorders (lupus, polyarteritis)
    2. History of cancer requiring chemotherapy and/or radiation
    3. Untreated hyperlipidemia
    4. Diabetes
    5. Ongoing active infection such as HIV, tuberculosis, sarcoidosis
    6. History of chronic transfusion
    7. Chronic renal failure/Dialysis
    8. Chronic lung disease characterized by need for oxygen
    9. Morbid obesity (weight >115 kg)
    10. Heart disease: history of congestive heart failure, history of severe coronary artery disease characterized by angioplasty or surgery, or history of angina
    11. Active hepatitis or liver failure
    12. Acquired or congenital immune deficiency
    13. History of psychoses (delusions, hallucinations) and/or schizophrenia
    14. Neurodegenerative disorders
    15. Genetic disorder associated with neurocognitive dysfunction such as Down Syndrome
    16. Other chronic illness or disorder other than SCD that will adversely affect the subject's performance in the study
14. Currently on Procrit or related drug that stimulates red blood cell production

Individuals who meet any of the following criteria are disqualified from enrollment as community controls in to the study:

1. Hb electrophoresis other than AA
2. Abnormal Hb (females: < 12 g/dL; males: < 13.5 g/dL)
3. Overt stroke
4. Previous abnormal MRI or CT
5. History of head injury that resulted in neurological symptoms or medical visit
6. Abnormal neurologic exam with focal findings
7. Mini-Mental Status Examination (MMSE) score of < 20
8. Profile of Mood States (POMS) score on the Depression-Dejection Subscale suggestive of a clinical depression (score > 40)
9. Alcohol consumption exceeding 14 drinks/week if female, 21 drinks/week if male
10. Drug abuse, defined as using non-prescribed medication
11. History of claustrophobia and/or presence of metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body
12. Pregnancy
13. Baseline blood pressure > 140/90 on two repeated measurements. A second measurement is needed only if the first is > 140/90
14. History of uncontrolled hypertension
15. Any chronic disorder that may result in neurocognitive or brain dysfunction including:

    1. Inflammatory arterial disorders (lupus, polyarteritis)
    2. History of cancer requiring chemotherapy and/or radiation
    3. Untreated hyperlipidemia
    4. Diabetes
    5. Ongoing active infection such as HIV, tuberculosis, sarcoidosis
    6. History of chronic transfusion
    7. Chronic renal failure/Dialysis
    8. Chronic lung disease characterized by need for oxygen
    9. Morbid obesity (weight > 115 kg)
    10. Heart disease: history of congestive heart failure, history of severe coronary artery disease characterized by angioplasty or surgery, or history of angina
    11. Active hepatitis or liver failure
    12. Acquired or congenital immune deficiency
    13. History of psychoses (delusions, hallucinations) and/or schizophrenia
    14. Neurodegenerative disorders
    15. Genetic disorder associated with neurocognitive dysfunction such as Down Syndrome
    16. Other chronic illness or disorder that will adversely affect the subject's performance in the study
16. Currently on Procrit or related drug that stimulates red blood cell production

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 212 participants, 160 will have sickle cell anemia, 52 will be matched controls based on gender, age, and education level
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Vichinsky, MD, Principal Investigator — Northern California CSCC (Children's Hospital Oakland)
Locations (12):
- United States (12):
  - University of Southern California, Los Angeles, California
  - Children's Hospital & Research Center at Oakland, Oakland, California
  - Memorial Cancer Institute, Hollywood, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Children's Medical Center at Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with HB SS/SB0 were recruited from 12 sickle cell centers from Dec 2004 through May 2008. To eliminate selection bias, all eligible patients at these centers were approached. Matched peer controls of African descent were recruited from patients' community-based churches or neighborhoods, and matched for gender, age and education.
Pre-assignment Details: The NP Battery and the MRI could be scheduled in either order. A 4 week visit window was set between screening and the first of the two procedures. An additional 4 week window was set between the first procedure and the second.
Groups:
- Phase I: Cases: These are patients diagnosed with sickle cell disease (confirmed by hemoglobin electrophoresis).
- Phase I: Controls: These are patients that do not have sickle cell disease (confirmed by hemoglobin electrophoresis); matched to cases by age, gender, and education level
Period: Overall Study
Arm/Group | Phase I: Cases | Phase I: Controls
Started | 160 | 52
Completed | 133 | 41
Not Completed | 27 | 11
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 11 | 5
Not completed — Lost to Follow-up | 15 | 4
Not completed — Administrative Reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Cases | Phase I: Controls | Total
Number analyzed (Participants) | 160 | 52 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 160 | 52 | 212
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.57 (8.95) | 33.10 (10.06) | 31.94 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 27 | 127
  Male | 60 | 25 | 85
Region of Enrollment [Number; unit: participants]
  United States | 160 | 52 | 212

OUTCOME MEASURES:

1. Primary Outcome: Wechsler Adult Intelligence Scale (WAIS)-III Performance IQ
Description: Extent of neurocognitive dysfunction in neurologically asymptomatic adult patients with sickle cell disease as measured by WAIS-III performance IQ. This quotient is based on an average of 100, with a standard deviation of 15. The Wechsler intelligence scales are not considered adequate measures of extremely high and low intelligence (IQ scores above 160 and below 40, respectively). The performance IQ is derived from scores on seven subtests: picture completion, picture arrangement, block design, object assembly, digit symbol, matrix reasoning, and symbol search.
Time Frame: Within 2 months of signing informed consent.
Population: Per protocol, no imputation used.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Phase I: Cases | Phase I: Controls
Number analyzed (Participants) | 144 | 45
Points on a scale | 90.6 (12.70) | 95.9 (12.13)
Statistical Analysis 1: Comparison: Phase I: Cases vs Phase I: Controls; Null hypothesis is no difference between cases and controls in the WAIS-III Perormance IQ (PIQ) Index. A linear model controlling for gender, age, and education was used to compare controls versus cases using an F statistic. Based on sample-size calculations, 120 patients and 36 controls were needed to have 80% power to detect an 8-point difference on the WAIS-III PIQ Index; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Adjusted for gender, age, and education; Mean Difference (Final Values) = -5.5, Standard Error of Mean 2.07 — Cases are lower than controls

2. Secondary Outcome: Participants With Brain Lacunae as Measured by Clinical MRI
Description: Particpants with imaging abnormalities as measured by MRI (Magnetic Resonance Imaging) specifically brain lacunae. Lacunar infarcts are 3-15 mm in diameter located at the basal ganglia, capsular and thalamic regions. Lesions located at the level of the anterior commisure are considered perivascular spaces unless >5 mm in diameter.
Time Frame: Within 2 months of informed consent
Population: Per protocol, no imputation.
Measure: Number; unit: Participants
Arm/Group | Phase I: Cases | Phase I: Controls
Number analyzed (Participants) | 144 | 45
Participants | 19 | 1
Statistical Analysis 1: Comparison: Phase I: Cases vs Phase I: Controls; Null hypothesis is no difference between cases and controls in the proportion of subjects with lacunae. This was tested using a Fisher's Exact Test; Test type: Superiority or Other; p = 0.048, Fisher Exact; Difference in proportions = .11, 95% CI [.026 to .199]

3. Secondary Outcome: Volume of Total Cortical Gray Matter as Measured by Volumetric MRI.
Description: The cortical gray matter is the gray matter of the cerebral cortex only and does not include subcortical gray matter such as hippocampus or basal ganglia.
Time Frame: Within 2 months of informed consent
Population: Per protocol, no imputations.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Phase I: Cases | Phase I: Controls
Number analyzed (Participants) | 144 | 45
mL | 543.5 (52.71) | 569.7 (63.04)

ADVERSE EVENTS:
Description: No adverse events or serious adverse events were reported or collected.
Arm/Group | Phase I: Cases | Phase I: Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
As a cross-sectional study, follow-up of patients not included. Age range of cases and controls not weighted enough to include elder population. Functional or perfusion brain measures not included. Biologic and genetic risk factors not included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No